CLINICAL TRIAL: NCT02141971
Title: Down Syndrome Biomarker Initiative: A Natural History Study of Alzheimer's Disease in Down Syndrome (Pilot Study)
Brief Title: Down Syndrome Biomarker Initiative (DSBI)
Acronym: DSBI
Status: Completed | Type: Observational
Sponsor: Michael Rafii (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Michael Rafii, Associate Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: DSBI
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Down Syndrome; Alzheimer's Disease
Keywords: Down syndrome; Alzheimer's disease; biomarkers; amyloid; tau
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-demented; Ages 30-40: Four non-demented Down syndrome patients between the ages of 30-40 years old
- Non-demented; Ages 40-50: Four non-demented Down syndrome patients between the ages of 40-50 years old
- Demented; Ages 50-60: Four demented Down syndrome patients between the ages of 50-60 years old

SUMMARY:
Non-randomized natural history study involving 12 subjects with Down Syndrome, who are aged 30-60 years old. This study will observe 3 different groups: four non-demented subjects between ages 30-40 years old, four non-demented subjects between ages 40-50 years old, and four demented subjects 50-60 years old.

Currently available longitudinal data in DS suggest a high rate of transition to dementia from the late 40s through the early 50s of these individuals. This, together with the universal presence of plaques in DS by their mid 40s makes this age range ideal for studying the development of AD.

DETAILED DESCRIPTION:
The overall goal of this project is to determine the relationships among the clinical, cognitive, imaging, genetic and biochemical biomarker characteristics of the entire spectrum of Alzheimer's disease (AD), as the pathology evolves from normal aging through very mild symptoms, to mild cognitive impairment (MCI), to dementia in adults with Down syndrome. This is a pilot study modeled after the Alzheimer's Disease Neuroimaging Initiative (ADNI) to inform the neuroscience community of AD in DS, identify diagnostic and prognostic markers, identify outcome measures that can be used in clinical trials, and help develop the most effective clinical trial scenarios.

AD is the most common dementia in humans and over the next decades will account for a major and increasing morbidity and mortality in the US and worldwide. AD is usually a sporadic disease and the commonly accepted hypothesis as to its etiology is the amyloid cascade hypothesis. There is tremendous activity in the pharmaceutical industry and academia directed towards development of disease modifying treatments, most commonly targeting amyloid, but also tau and other mechanisms. Most efforts are directed towards Mild to Moderate AD or prodromal AD with relatively little work on prevention of AD due to various challenges, including identification of healthy people who would be treated.

Down syndrome is the most common chromosomal disorder in humans, caused by triplication of chromosome 21, accounting for ~1/740 live births in the USA even with routine prenatal screening. In addition to mental retardation and the other classical signs of DS, 100% of people with DS will develop the pathological hallmarks of AD (plaques and tangles) by their 40s and ~80% of people with DS will eventually develop clinical dementia. The primary cause is the triplication of the APP gene on chromosome 21, resulting in 50% greater levels of both APP mRNA and protein. That the disease in DS is indeed AD is supported by pathological, molecular, in-vitro, biomarker and clinical evidence.

People with DS have been followed at major centers in the US and EU for decades with large amounts of clinical and psychometric data gathered and analyzed. There is, however, very little data on CSF biomarkers due to the difficulty of performing lumbar punctures in DS subjects. Only recently has data begun to be gathered from imaging modalities, including Amyloid imaging.

There is no gold standard for the diagnosis of AD in this population and, due to the MR, the standard instruments cannot be used. Most major centers have developed specific instruments that can follow cognitive and functional performance and allow the detection of dementia. The data gathered over the past decades allows the construction of a curve describing the transition to dementia in this population and shows the transition beginning in the mid 40s with a steep slope around the age of 50.

DS is, in effect, a population highly enriched for people who will, with a very high probability develop AD, and it is expected that only with an ADNI-like study can the investigators better understand the trajectory of transition to dementia in this population.

The ultimate goal of this project is to develop treatments for the prevention of AD in this population. Because if the investigators would know at what age the slope of transition to dementia is steepest, a study could be done in a specific age range and require much fewer subjects and time and expense than a study in the general population (where it is currently impossible to determine which healthy individuals will likely develop dementia over the next few years and even if there were, thousands would have to be screened to ID these few). A study in the general population might need to enroll tens of thousands of subjects to observe sufficient transitions to dementia. The investigators estimate that such a study in DS would require about 170 subjects per arm for a 36 month study. Success in such a study would provide the confidence to commit the resources for a larger study in the general population.

As mentioned above, there is minimal CSF data and imaging is only beginning. Thus biomarkers for AD in DS are less developed than in the general population. Additional biomarkers could be helpful in studying AD in DS. A biomarker that could increase the ability to predict transition to dementia in an individual (as opposed to the investigators current ability on a population level) would increase the efficiency of any study. The ability to track the progression or improvement of dementia might also be useful. If a biomarker indicated transition to dementia earlier than any clinical instrument, a prevention study could conceivably be conducted at younger ages with greater chance of success. In addition to DS, such a biomarker would also be useful in the general population.

This study is a pilot study for a larger scale biomarker study which, as described, would enable better understanding of biomarkers and the natural history of AD in DS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 30 to 60 years of age inclusive with chromosome karyotype of Down Syndrome due to Trisomy 21.
* Subjects must have a study partner (parent or other reliable caregiver) who has at least 10 hours of contact and who agrees to accompany the subject to all clinic visits and provide information about the subject's behavior and symptoms.
* Participant is able to speak/communicate.
* Subject is willing and has no contraindications to MRI scanning.
* Participant or parent/legal guardian provides consent.
* Participant must agree to allow for indefinite storage of his/her data and samples.

Exclusion Criteria:

* Patients who are anarthric or mute.
* Patients who do not meet the criteria for the diagnosis of DS.
* Patients unwilling or unable to participate in all tests and procedures.
* Unstable medical or behavioral issues.
* Unable or unwilling to perform MRI and/or PET imaging.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of decline as measured by cognitive, functional and behavioral tests | 3 years

SECONDARY OUTCOMES:
Rate of conversion will be evaluated among all age groups | 3 years
Rate of volume change of whole brain, hippocampus, and other structural Magnetic resonance imaging (MRI) measures. | 3 years
Rates of change on each specified biochemical biomarkers | 3 years
Rates of change of glucose metabolism as measured by fluorodeoxyglucose positron emission tomography (FDG-PET) imaging | 2 years
Extent of amyloid deposition as measured amyloid PET imaging | 3 years
Rates of change on retinal amyloid measures. | 3 years
Correlations among biomarkers and cognitive change. | 3 years
Correlations of Tau deposition as measured by 18F-AV-1451 PET (Tau) imaging with other biomarkers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Rafii, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonsson T, Atwal JK, Steinberg S, Snaedal J, Jonsson PV, Bjornsson S, Stefansson H, Sulem P, Gudbjartsson D, Maloney J, Hoyte K, Gustafson A, Liu Y, Lu Y, Bhangale T, Graham RR, Huttenlocher J, Bjornsdottir G, Andreassen OA, Jonsson EG, Palotie A, Behrens TW, Magnusson OT, Kong A, Thorsteinsdottir U, Watts RJ, Stefansson K. A mutation in APP protects against Alzheimer's disease and age-related cognitive decline. Nature. 2012 Aug 2;488(7409):96-9. doi: 10.1038/nature11283. PMID 22801501
- [Background] Netzer WJ, Powell C, Nong Y, Blundell J, Wong L, Duff K, Flajolet M, Greengard P. Lowering beta-amyloid levels rescues learning and memory in a Down syndrome mouse model. PLoS One. 2010 Jun 3;5(6):e10943. doi: 10.1371/journal.pone.0010943. PMID 20532168
- [Background] Roe CM, Mintun MA, Ghoshal N, Williams MM, Grant EA, Marcus DS, Morris JC. Alzheimer disease identification using amyloid imaging and reserve variables: proof of concept. Neurology. 2010 Jul 6;75(1):42-8. doi: 10.1212/WNL.0b013e3181e620f4. PMID 20603484
- [Background] Zigman WB, Lott IT. Alzheimer's disease in Down syndrome: neurobiology and risk. Ment Retard Dev Disabil Res Rev. 2007;13(3):237-46. doi: 10.1002/mrdd.20163. PMID 17910085
- [Derived] Rafii MS, Wishnek H, Brewer JB, Donohue MC, Ness S, Mobley WC, Aisen PS, Rissman RA. The down syndrome biomarker initiative (DSBI) pilot: proof of concept for deep phenotyping of Alzheimer's disease biomarkers in down syndrome. Front Behav Neurosci. 2015 Sep 14;9:239. doi: 10.3389/fnbeh.2015.00239. eCollection 2015. PMID 26441570
- See also: Related Info — http://downsyndrome.ucsd.edu